CLINICAL TRIAL: NCT00078130
Title: Bup/Nx - Facilitated Rehab for Opioid Dependent Adolescents
Brief Title: Buprenorphine/Naloxone - Facilitated Rehabilitation for Opioid Dependent Adolescents - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: George Woody, M.D., University of Pennsylvania
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-CTN-0010-1
Record Dates: First submitted 2004-02-19; First posted 2004-02-20 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Opioid-Related Disorders
Keywords: opioid dependence; behavioral intervention
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
The purpose of this study is to compare two 3-month treatments for adolescents/young adults who are addicted to heroin: buprenorphine/naloxone combined with psychosocial therapy and treatment as usual, a 7-14 day detoxification with buprenorphine and three weeks of psychosocial therapy.

ELIGIBILITY:
Male and non-pregnant female subjects seeking outpatient treatment for opioid dependence with physiological features without serious medical or psychiatric disorders.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 223
Dates: Start 2003-07; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Opiate abstinence

CONTACTS AND LOCATIONS:
Overall Officials: George Woody, M.D., Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Mercy Hospital, Portland, Maine
  - Mountain Manor, Baltimore, Maryland
  - ASAP, Albuquerque, New Mexico
  - Duke Addictions Program, Durham, North Carolina

REFERENCES:
- [Derived] Nielsen S, Tse WC, Larance B. Opioid agonist treatment for people who are dependent on pharmaceutical opioids. Cochrane Database Syst Rev. 2022 Sep 5;9(9):CD011117. doi: 10.1002/14651858.CD011117.pub3. PMID 36063082
- [Derived] Schackman BR, Leff JA, Polsky D, Moore BA, Fiellin DA. Cost-effectiveness of long-term outpatient buprenorphine-naloxone treatment for opioid dependence in primary care. J Gen Intern Med. 2012 Jun;27(6):669-76. doi: 10.1007/s11606-011-1962-8. Epub 2012 Jan 4. PMID 22215271
- [Derived] Subramaniam GA, Warden D, Minhajuddin A, Fishman MJ, Stitzer ML, Adinoff B, Trivedi M, Weiss R, Potter J, Poole SA, Woody GE. Predictors of abstinence: National Institute of Drug Abuse multisite buprenorphine/naloxone treatment trial in opioid-dependent youth. J Am Acad Child Adolesc Psychiatry. 2011 Nov;50(11):1120-8. doi: 10.1016/j.jaac.2011.07.010. PMID 22024000
- [Derived] Polsky D, Glick HA, Yang J, Subramaniam GA, Poole SA, Woody GE. Cost-effectiveness of extended buprenorphine-naloxone treatment for opioid-dependent youth: data from a randomized trial. Addiction. 2010 Sep;105(9):1616-24. doi: 10.1111/j.1360-0443.2010.03001.x. Epub 2010 Jul 12. PMID 20626379
- [Derived] Meade CS, Weiss RD, Fitzmaurice GM, Poole SA, Subramaniam GA, Patkar AA, Connery HS, Woody GE. HIV risk behavior in treatment-seeking opioid-dependent youth: results from a NIDA clinical trials network multisite study. J Acquir Immune Defic Syndr. 2010 Sep;55(1):65-72. doi: 10.1097/QAI.0b013e3181d916db. PMID 20393347
- [Derived] Chakrabarti A, Woody GE, Griffin ML, Subramaniam G, Weiss RD. Predictors of buprenorphine-naloxone dosing in a 12-week treatment trial for opioid-dependent youth: secondary analyses from a NIDA Clinical Trials Network study. Drug Alcohol Depend. 2010 Mar 1;107(2-3):253-6. doi: 10.1016/j.drugalcdep.2009.10.014. Epub 2009 Nov 30. PMID 19948382
- [Derived] Woody GE, Poole SA, Subramaniam G, Dugosh K, Bogenschutz M, Abbott P, Patkar A, Publicker M, McCain K, Potter JS, Forman R, Vetter V, McNicholas L, Blaine J, Lynch KG, Fudala P. Extended vs short-term buprenorphine-naloxone for treatment of opioid-addicted youth: a randomized trial. JAMA. 2008 Nov 5;300(17):2003-11. doi: 10.1001/jama.2008.574. PMID 18984887